CLINICAL TRIAL: NCT03831620
Title: The Crosstalk Between Calcium-sensing Receptor Signaling and Endocannabinoid System in Primary Hyperparathyroidism
Acronym: Targeting CaSR
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-02218
Record Dates: First submitted 2019-01-25; First posted 2019-02-06 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Primary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite the strong association of hyperparathyroidism with arachidonic acid related lipid signals, little research has been performed over the years. A better understanding of the link between arachidonic acid remodeling, prostaglandin and endocannabinoid production with primary hyperparathyroidism in primary tissue/cells might open up new avenues for biomarker and thus to a potential therapeutic target.

Arachidonic acid remodeling might also have an impact on depression and elevated cytokines in patients with primary hyperparathyroidism. The investigators therefore will assess the correlation between postoperative improvement of PHQ-9 and cytokine levels with arachidonic acid remodeling.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Primary hyperparathyroidism with planned surgery
* Written informed consent

Exclusion Criteria:

* Age <18 years
* Secondary/tertiary hyperparathyroidism
* Renal insufficiency
* Participant is pregnant
* Participant is incapable of giving an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary hyperparathyroidism with planned surgery
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Activity-based protein profiling (ABPP) will be used to assess the enzymes involved in calcium induced stress signals and endocannabinoid activation | 2 months

SECONDARY OUTCOMES:
Measurement of the level of parathyroid hormone | 2 months
Measurement of the level of calcium | 2 months
Measurement of the level of cortisol | 2 months
Measurement of the level of 25-hydroxyvitamin D | 2 months
Measurement of the levels of the enzymes involved in the endocannabinoid system activation (diacylglycerol lipase; monoacylglycerol lipase, phospholipases, cyclooxygenases) | 2 months
Measurement of the level of endocannabinoids, arachidonic acid species, prostanoids and related anti-inflammatory lipids | 2 months
Measurement of the level of IL-6 and TNF-α | 2 months
Assessment of Patient Health Questionnaire - 9 | 2 months
  The Patient Health Questionnaire (PHQ-9) is described as a valid depression scale with good sensitivity and specificity for detecting depressive disorders, ranging from 1 to 27.
  Depression severity:
  1 to 4: minimal; 5 to 9: mild; 10 to 14: moderate; 15 to 19: moderately severe; 20 to 27: severe

CONTACTS AND LOCATIONS:
Overall Officials: Reto Kaderli, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Department of visceral surgery and transplant surgery, Berne University Hospital, Bern, Switzerland